CLINICAL TRIAL: NCT02114970
Title: Comparing Paper-based and Tablet-delivered Informed Consent for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Nimali Jayasinghe, Assistant Professor, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1401014708
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Tablet-delivered Informed Consent; Paper-based Informed Consent
Keywords: Older Adults; Informed Consent; Technology; Tablet-delivered

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Focus Group- paper and tablet consent (Other): Participation in a focus group of other older adults, lasting 120 minutes. Participants will answer semi-structured questions in a group format, describing their impressions of both a prototype tablet-delivered and a paper consent.
  Interventions: Other: Focus Group- paper and tablet consent
- Randomized- paper consent (Active Comparator): Participants will review a mock paper consent form with a study clinician, and complete a series of questionnaires assessing their comprehension of material covered and general experience with the paper informed consent form.
  Interventions: Other: Randomized- paper consent
- Randomized- Tablet-delivered consent (Active Comparator): Participants will review a mock tablet-delivered consent form with a study clinician, and complete a series of questionnaires assessing their comprehension of material covered and general experience with the tablet-delivered informed consent.
  Interventions: Other: Randomized- Tablet-delivered consent

INTERVENTIONS:
Other: Randomized- paper consent
  Arms: Randomized- paper consent
Other: Randomized- Tablet-delivered consent
  Arms: Randomized- Tablet-delivered consent
Other: Focus Group- paper and tablet consent
  Arms: Focus Group- paper and tablet consent

SUMMARY:
The investigators will develop and test a tablet-delivered informed consent process. In a preliminary phase of the study, older adults will provide feedback on a prototype tablet-delivered consent by participating in a focus group. In a separate second phase, older adults will be randomly assigned to a tablet-delivered or paper-delivered consent condition in which their comprehension of material covered in the consent will be assessed.

DETAILED DESCRIPTION:
Clinical research is crucial for advancing healthcare, but patients must be able to make informed and voluntary choices about whether or not to participate in a research study. The informed consent process aspires to convey the purpose of research, the procedures involved, and the potential harms and benefits of taking part. Yet, the challenge of making informed consent easy to follow and understand is great: there are specific challenges for older research populations.

This study will develop and test a tablet-delivered informed consent process. The study will have two phases.

In the first phase, focus groups comprised of older adults will give their impressions of both a prototype tablet-delivered and paper consent, and the prototype will be refined according to feedback.

The second phase will evaluate whether older subjects judge a tablet-delivered consent to be more user-friendly than a paper-based version. It will also evaluate whether older subjects who participate in a tablet-delivered consent process have a better understanding of the research than those who participate in the paper-based version, and whether they remember the research details more fully after a one-week delay.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Cognitively intact
* Ability to speak and read English

Exclusion Criteria:

* Legal blindness
* Severe hearing loss not corrected by assistive device
* Inability to use hands to swipe a tablet's touch screen
* No working telephone in the home

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
University of California San Diego Brief Assessment of Capacity to Consent (UBACC) | immediately following intervention

SECONDARY OUTCOMES:
study-specific measure of user-friendliness consent process | immediately following intervention
UBACC | One week following intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nimali Jayasinghe, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States